CLINICAL TRIAL: NCT06321640
Title: POSITive: Prospective Observational Study for the Multidimensional Analyses of Resistance and Toxicity to Immune- and Targeted-therapies
Brief Title: Study for the Multidimensional Analyses of Resistance and Toxicity to Immune- and Targeted-therapies.
Acronym: POSITive
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1777
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Lung Cancer; Melanoma; Head and Neck Cancer; Urothelial Carcinoma; Colorectal Cancer; Liver Metastases; Lung Metastases
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Melanoma; Head and Neck Neoplasms; Carcinoma, Transitional Cell; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A surgical specimen will be collected. The sample will be processed regularly for diagnostic histopathology.One additional tumor specimen beyond the diagnostic biopsy will be collected using a single-pass technique. If a single additional specimen is collected, it will be processed in formalin according to the standard pathology procedure.Peripheral blood (18 ml in total) and Bone Marrow Aspirate (10 ml) will be collected.A biological specimen relevant for the toxic event will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cohort A: primarily operable disease, candidate to adjuvant: This cohort includes any patient with nonmetastatic disease, candidate to surgery as primary treatment, for whom adjuvant therapy with targeted or immune therapy is recommended based on prior information obtained on the diagnostic biopsy. This cohort represents a control group, for whom high-throughput DNA/RNA sequencing is considered feasible in the vast majority of cases, and will not be considered in the computation of the primary endpoint. Small groups representative of relevant diseases will be collected, as follows:
  * Breast
  * Lung
  * Melanoma
  * Head and Neck
  * Urothelial
  * Colorectal cancer
  * Metastasectomy from lung or liver, from any cancer
  Interventions: Genetic: Cohort A: primarily operable disease, candidate to adjuvant
- Cohort B: locally advanced disease: Patients in this cohort are eligible if diagnosed with or highly suspected of locally advanced (nonmetastatic) neoplasm and candidate to a diagnostic/confirmatory biopsy and subsequent treatment with targeted therapy, immune therapy or radiotherapy, where the treatment is administered with potentially curative intent. Patients in this cohort may be considered for enrolment prior to a formal diagnosis, so the study should be offered on the basis of a high suspicion of invasive cancer upon radiological evidence.Cohort B1: patients who, at the moment of biopsy, are expected to be subsequently treated with targeted therapy. Cohort B2: patients who, at the moment of biopsy, are expected to be subsequently treated with immune therapy. Cohort B3: patients who, at the moment of biopsy, are expected to be treated with combined chemo-immuno-radiotherapy
  Interventions: Genetic: Cohort B: locally advanced disease
- Cohort C: metastatic disease: In this cohort, patients are eligible if diagnosed with invasive cancer with radiologically proven metastatic localization and candidate to treatment with targeted or immune therapy.
  Cohort C1: patients candidate to targeted therapy Cohort C2: patients candidate to immune therapy
  Interventions: Genetic: Cohort C: metastatic disease
- Cohort D: Progressive disease: In this cohort, patients are eligible if a tumor biopsy is considered indicated by the referring physician upon disease progression to prior treatment in the metastatic setting or for hematological neoplasms. Definition of progression is based on the investigator's judgement and does not strictly require RECIST 1.1 definition, although all relevant radiological data will be collected whenever possible. Tumor biopsy must be collected no more than 6 months after the documented date of progression.
  Subgroups include: Cohort D1: progression disease to targeted. Patients whose last treatment at the moment of enrolment is a targeted agent.
  Cohort D2: progression disease to immune. Patients whose last treatment at the moment of enrolment is an immunotherapeutic agent Cohort D3: potential off-label treatment. Any patient that has exhausted standard treatment and that in the judgement of the investigator may benefit from an exome-wide mutational screen to identify actionable alterations
  Interventions: Genetic: Cohort D: Progressive disease
- Cohort E: Hematological neoplasms: Cohort E1: Any patient that is expected to be treated with targeted agents. Special consideration will be given to patients affected by chronic lymphoid leukemia and follicular lymphoma treated with Bruton´s tyrosine kinase (BTK) inhibitor, Phosphoinositide 3-kinase inhibitor, B-cell lymphoma 2 inhibitor +/- monoclonal antibodies.
  Cohort E2: Any patient that is expected to be treated with immunotherapy. Special consideration will be given to patients affected by Hodgkin lymphoma and Diffuse Large B-cell lymphoma treated with Immune checkpoint inhibitors, Tafasitamab/Lenalidomide, immunoconjugates.
  Interventions: Genetic: Cohort E: Hematological neoplasms
- Cohort F: Toxicity: In this cohort, patients are enrolled upon experiencing an adverse event of grade 3/4 as per Common Terminology Criteria for Adverse Events version 5.0 that, in the opinion of the investigator, is unequivocally caused by a targeted or immune therapeutic. The event may occur at any time after the last dose of the drug. Events may be of any nature but particular attention will be given to those events for which pathophysiology is currently poorly understood.Cohort F1: toxicity to Targeted therapy. Patients experiencing Grade 3-Grade 4 adverse events due to targeted therapy Cohort F2: toxicity to Immune therapy. Patients experiencing Grade 3-Grade 4 adverse events due to Immune therapy.
  Interventions: Genetic: Cohort F: Toxicity

INTERVENTIONS:
Genetic: Cohort A: primarily operable disease, candidate to adjuvant — This cohort includes any patient with nonmetastatic disease, candidate to surgery as primary treatment, for whom adjuvant therapy with targeted or immune therapy is recommended based on prior information obtained on the diagnostic biopsy. This cohort represents a control group, for whom high-throughput DNA/RNA sequencing is considered feasible in the vast majority of cases, and will not be considered in the computation of the primary endpoint
  Groups: Cohort A: primarily operable disease, candidate to adjuvant
Genetic: Cohort B: locally advanced disease — Patients in this cohort are eligible if diagnosed with or highly suspected of locally advanced (nonmetastatic) neoplasm and candidate to a diagnostic/confirmatory biopsy and subsequent treatment with targeted therapy, immune therapy or radiotherapy, where the treatment is administered with potentially curative intent. Patients in this cohort may be considered for enrolment prior to a formal diagnosis, so the study should be offered on the basis of a high suspicion of invasive cancer upon radiological evidence.
  Groups: Cohort B: locally advanced disease
Genetic: Cohort C: metastatic disease — In this cohort, patients are eligible if diagnosed with invasive cancer with radiologically proven metastatic localization and candidate to treatment with targeted or immune therapy.
  Groups: Cohort C: metastatic disease
Genetic: Cohort D: Progressive disease — In this cohort, patients are eligible if a tumor biopsy is considered indicated by the referring physician upon disease progression to prior treatment in the metastatic setting or for hematological neoplasms. Definition of progression is based on the investigator's judgement and does not strictly require RECIST 1.1 definition, although all relevant radiological data will be collected whenever possible. Tumor biopsy must be collected no more than 6 months after the documented date of progression.
  Groups: Cohort D: Progressive disease
Genetic: Cohort E: Hematological neoplasms — Any patient that is expected to be treated with targeted agents. Special consideration will be given to patients affected by chronic lymphoid leukemia and follicular lymphoma treated with BTKi, PI3Ki, BCL-2i +/- monoclonal antibodies. Any patient that is expected to be treated with immunotherapy. Special consideration will be given to patients affected by Hodgkin lymphoma and Diffuse Large B-cell lymphoma treated with ICIs, Tafasitamab/Lenalidomide, immunoconjugates.
  Groups: Cohort E: Hematological neoplasms
Genetic: Cohort F: Toxicity — In this cohort, patients are enrolled upon experiencing an adverse event of grade 3/4 as per CTCAE v 5.0 that, in the opinion of the investigator, is unequivocally caused by a targeted or immune therapeutic. The event may occur at any time after the last dose of the drug. Events may be of any nature but particular attention will be given to those events for which pathophysiology is currently poorly understood (severe myocardial or neurologic Immune-related events or DS-8201-induced pneumonitis)
  Groups: Cohort F: Toxicity

SUMMARY:
Novel treatment modalities like targeted therapies and Immune checkpoint inhibitors have revolutionised the therapeutic landscape in oncology and hematology, significantly improving outcomes even in clinical contexts in which little improvement had been observed for decades such as metastatic melanoma, lung cancer, and lymphoproliferative neoplasms such as chronic lymphoid leukemia or Hodgkin lymphoma. However, major issues remain unsolved, given the frequent occurrence of primary or secondary resistance and the still incomplete understanding of the physiopathology of adverse events, which represent a major cause of morbidity and treatment interruption and often remain difficult to treat and diagnose. In this complex landscape, identifying the best treatment option for each patient remains challenging. For both targeted therapies and Immune checkpoint inhibitors, several biomarkers have been reported, but their implementation in clinical practice is still uncommon, and most of the decision-making process remains based on purely clinical considerations or constraints dictated by the regulatory bodies. Obstacles to biomarker-driven decision making are manifold and include insufficient understanding of the underlying biology, lack of strong evidence on their predictive power and limited tumor sampling, which may be circumvented by non-invasive techniques such as liquid biopsies.

DETAILED DESCRIPTION:
Biomarkers to predict response and toxicity to Targeted Therapies. Targeted therapies such as kinase inhibitors are usually associated with extremely elevated response rates, precisely because their use requires the prior detection of a companion biomarker. However, secondary resistance almost invariably develops, resulting in often moderate improvements in overall survival despite major delays in disease progression. Resistance mechanisms can be broadly classified in two groups: i) "cis"-mutations that directly impinge on the binding of the drug to its target and ii) "trans" alterations that activate additional pathways able to override drug-induced inhibition or transcriptional upregulation of parallel pathways . In both cases these mutations are mostly acquired as an evolutionary response to the selective environment generated by the drug itself, and their identification is crucial to identify potential subsequent treatments able to circumvent the resistance mechanism. As more targeted therapies enter clinical practice, including novel classes like Antibody-drug conjugates (which maintain high target specificity but have completely different mechanisms of action), extensive investigation of the molecular mechanisms associated with secondary resistance becomes more and more relevant.

Furthermore, many targeted therapies are associated with specific toxicities such as interstitial lung disease that are themselves poorly characterized from a mechanistic point of view, and this lack of knowledge prevents effective diagnosis and treatment.

Biomarkers to predict response and toxicity to Immune Checkpoint Inhibitors. Several biomarkers with predictive power in Immune checkpoint inhibitorsI-treated patients have been reported (e.g. tumor mutational burden, extent of tumour T-cell infiltration at baseline, expression by tumor cells of the respective Immune checkpoint inhibitors targets). However each of these, individually, bears very little accuracy for outcome . A recent meta-analysis of tumor-intrinsic data across >1,000 patients and multiple tumor types elaborated a multivariable predictive model for each cancer type using 11 features derived from genomic (whole exome sequencing ) and transcriptomic (total ribonucleic acid sequencing ) data of primary tumors (see below for the list of markers). The multivariable predictor attained an Afea Under the Receiver-Operating Characteristic value of 0.86, thus strongly indicating that an integrated assessment of multiple and novel biomarkers achieves an accuracy that can significantly impact on decision making. Moreover, recent findings suggest a critical role for the gut microbiome. Notably, specific species in the gut microbiota promote anti-cancer immunity during Immune checkpoint inhibitors treatment, which can be transferred by faecal microbiome transplantation to rescues Immune checkpoint inhibitors sensitivity in model systems . Underlying molecular mechanisms, however, are unknown, and may involve immunological mimicry of tumour neoantigens by microbial peptides from the gut or tumor microbiota .

The issue of drug-related toxicities (Immune-related Adverse events) is possibly even more crucial in Immune checkpoint inhibitors-treated patients. Immune-related Adverse events commonly develop after a long latency, are associated with significant morbidity and mortality and often represent a reason for treatment discontinuation and disease relapse. Immune-related Adverse events are often difficult to diagnose, since their pathophysiology is different from that of clinically similar idiopathic autoimmune disorders. Despite the definition of consensus guidelines on the diagnosis and treatment of Immune-related Adverse events, therapeutic options are limited and invariably include generalized immune suppression, to the detriment of the anticancer response. Biomarkers strongly predictive or diagnostic of Immune-related Adverse events have not been identified to date. Some studies have identified specific cytokine combinations but these studies remain correlative and require validation in larger cohorts and different clinical contexts.

ELIGIBILITY:
Inclusion Criteria:

* age>18 yrs old
* histological diagnosis of any cancer
* signed informed consent
* fulfills criteria described in cohort definition
* Clinical indication for a diagnostic biopsy

Exclusion Criteria:

Performance Status (ECOG) >2

* life expectancy < 3 months
* unwilling to receive treatment at IEO for at least 6 months after enrolment
* active pregnancy at the moment of enrolment
* for cohort F: use of steroids (higher than 10 mg prednisone-equivalent) or other major immunosuppressive drug (e.g. tocilizumab) in the 14 days prior to the baseline sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with solid tumors
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in each cohort that will obtain a full "core" omic characterization. | 2 months
  For cohorts A-E:
  i) Whole Exome Sequencing of tumor samples (biopsy/surgery) ii) ribonucleic acid sequence iii) Whole-genome "shotgun" metagenomic sequencing of fecal samples
  For cohorts C and D:
  i) Computation of the 11-parameter multivariable score: clonal Tumor Mutation Load, indel Tumor Mutation Load, nonsense mediated decay-escape Tumor Mutation Load, tobacco signature etc.
  For cohorts E,F i) High throughput cytokine bead array on plasma samples ii) ribonucleic acid sequence iii) Whole-genome "shotgun" metagenomic sequencing of fecal samples

SECONDARY OUTCOMES:
Percentage of patients with complete clinical data collection over the expected follow-up time and with successful biobanking. | 2 years
  Percentage of patients with complete clinical and laboratory data collection over the expected follow-up time (2 years); Percentage of patients with successful biobanking (presence of at least 1 frozen tumor sample, 1 vial of EDTA blood, 2 vials of plasma at T0, T1, T2, 1 vial of feces at T0, T1, T2).Somatic mutations associated with sensitivity, primary/secondary resistance and toxicity;Prevalence of specific signaling-pathway transcriptional-activation signatures associated with sensitivity, primary/secondary resistance and toxicity;Prevalence of specific microbiota signatures associated with sensitivity, primary/secondary resistance and toxicity; Prevalence of germline variants associated with sensitivity, primary/secondary resistance and toxicity;

CONTACTS AND LOCATIONS:
Overall Officials: Luca Mazzarella, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of oncology, Milan, Italy